CLINICAL TRIAL: NCT03995004
Title: The Effect of Melatonin on Postoperative Pain Reduction After Orthognathic Surgery
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to secure study medication supply
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 19-221
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-10

CONDITIONS: Effect of Drugs
Keywords: melatonin; orthognathic; pain; surgery
MeSH Terms: conditions — Pain | interventions — Melatonin; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: M: Oral Melatonin 10mg / IV Normal Saline D: Placebo cap / IV Dexamethasone 4mg DM: Oral Melatonin 10mg / IV Dexamethasone 4mg
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical capsules for melatonin and placebo Clear fluid of the same volume for IV dexamethasone vs normal saline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Melatonin (Experimental): Oral Melatonin 10mg at night time one day before the surgery and on the surgical day, and continued at bedtime on the surgical day, post-surgery day 1 and day 2.
  IV Normal Saline (1mL) on induction and continued q12h for 4 more doses.
  Interventions: Drug: Melatonin
- Dexamethasone (Active Comparator): Placebo capsules at night time one day before the surgery and on the surgical day, and continued at bedtime on the surgical day, post-surgery day 1 and day 2.
  IV Dexamethasone 4mg/1mL on induction and continued q12h for 4 more doses
  Interventions: Drug: Dexamethasone Sodium Sulphate 4mg/1mL
- Dexa_Melatonin (Experimental): Oral Melatonin 10mg at night time one day before the surgery and on the surgical day, and continued at bedtime on the surgical day, post-surgery day 1 and day 2.
  IV Dexamethasone 4mg/1mL on induction and continued q12h for 4 more doses
  Interventions: Drug: Melatonin; Drug: Dexamethasone Sodium Sulphate 4mg/1mL

INTERVENTIONS:
Drug: Melatonin — Melatonin (N-acetyl-5-methoxytryptamine) is a neurohormone that is endogenously produced and secreted by the pineal gland in the brain following a circadian rhythm, with a plasma concentration highest at night and lowest during the day.
  Arms: Dexa_Melatonin; Melatonin
Drug: Dexamethasone Sodium Sulphate 4mg/1mL — Dexamethasone is a glucocorticoid commonly used in orthognathic surgery to reduce postoperative facial edema by its potent anti-inflammatory effect
  Other Names: Decadron
  Arms: Dexa_Melatonin; Dexamethasone

SUMMARY:
Orthognathic surgery is a procedure performed to correct dentofacial deformities. It involves osteotomy at the facial skeleton. Considerable pain is expected in the early recovery period.

Melatonin is a hormone that is produced naturally by the body. Synthetic Melatonin is available over the counter for the management of sleeping disorder and jetlag. Clinically, Melatonin can also be used to reduce pain and analgesic consumption in patients undergoing surgery.

Dexamethasone is a type of steroid. It can suppress the inflammatory response. It is an anti-inflammatory, anti-allergic drug. It is commonly used in head and neck and oral surgery for its anti-inflammatory effect to reduce swelling.

This study aims evaluate the efficacy of oral melatonin in the pain reduction following orthognathic surgery.

This is a double-blinded randomized controlled trial. We will recruit 87 patients who are scheduled for double-jaw orthognathic surgery to participate in this three-year study. The study lasts for 2 weeks. Participant will be randomly allocated by computer to one of the three groups. (1) Group D will receive dexamethasone only; (2) Group M will receive melatonin only; and (3) Group DM both melatonin and dexamethasone.

Postoperative pain level and perioperative plasma levels of inflammatory markers and anti-oxidizing enzymes will be recorded and compared among the study groups.

DETAILED DESCRIPTION:
Melatonin (N-acetyl-5-methoxytryptamine) is a neurohormone that is endogenously produced and secreted by the pineal gland in the brain following a circadian rhythm, with a plasma concentration highest at night and lowest during the day.

The normal physiological roles of melatonin in the human body are to regulate diurnal rhythm, sleep, mood, immunity, reproduction, intestinal motility, and metabolism. Oral supplemental melatonin has been used in the management of jetlag and other sleep disorders. Recently, melatonin's analgesic, antioxidative, and neuroprotective properties have been highlighted in a number of animal models and a few human trials, although the exact cellular mechanism is still not yet clearly established. In surgical human trials, some conflicting data have been presented regarding the analgesic properties of exogenous melatonin supplement. Whilst the large proportion of studies showed that perioperative administration of melatonin yielded significantly positive effects in the reduction of postsurgical pain, and the reduction of overall morphine consumption, others demonstrated the opposite with no significant effects in pain experience. The reason for this could be related to the dosage, route of administration, and/or time of administration. To date, there is still no consensus on a standardized dosing regimen for melatonin. In non-surgical trials, melatonin has shown promising benefits in many degenerative diseases and conditions related to chronic inflammation and oxidative stress. Amongst many, the reported positive effects of melatonin ranged from the reduction of radiation dermatitis, control of signs and symptoms of ulcerative colitis, management of chronic retinopathy, and reduction of lung oxidative stress in chronic obstructive pulmonary disease patients.

Hypothesis:

Melatonin can significantly reduce postoperative pain after orthognathic surgery. Antioxidative enzyme activity and level will be elevated and the level of inflammatory markers are reduced. Melatonin has a synergistic effect with dexamethasone.

This is a double-blinded randomized controlled trial. We will recruit 87 patients who are scheduled for double-jaw orthognathic surgery to participate in this three-year study. The study lasts for 2 weeks. Participant will be randomly allocated by computer to one of the three groups. (1) Group D will receive dexamethasone only; (2) Group M will receive melatonin only; and (3) Group DM both melatonin and dexamethasone.

Postoperative pain level and perioperative plasma levels of inflammatory markers and anti-oxidizing enzymes will be recorded and compared among the study groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class I
* Age between 18 - 60 inclusive

Exclusion Criteria:

* Pregnancy
* Any pre-existing systemic condition
* Previous history of orthognathic surgery
* Adverse reaction or allergic to oral melatonin
* Need for distraction osteogenesis
* Patient with chronic pain
* Patients with known psychological disorders
* Currently taking oral steroid or anti-inflammatory medication or any analgesic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Subjective pain perception | 14 days
  Self-reported pain level by numerical rating scale
Total analgesic consumption | 14 days
  Total amount of postoperative analgesic consumed

SECONDARY OUTCOMES:
Time to first analgesic | 1 day
  Time for patient to request for first dose of analgesic after the surgery (mins)
Plasma levels of melatonin | 16 days
  Plasma levels of melatonin (pg/mL)
Plasma levels of inflammatory markers | 16 days
  IL-6 and IL-10 (pg/mL)
Plasma levels of hydrogen peroxide | 16 days
  Plasma levels of hydrogen peroxide (µM)
Plasma levels and activities of antioxidative enzymes | 16 days
  superoxide dismutase (U/mL), catalase ((nmol/min/mL), and glutathione peroxidase (nmol/min/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Winnie WS CHOI, PhD, MDS, Principal Investigator — The University of Hong Kong
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No